CLINICAL TRIAL: NCT06641492
Title: A Randomized Controlled Trial Evaluating a Trans-Theoretical-Model-based Online Intervention Delivered by Fully-automated Chatbot in Increasing Physical Activity Among Inactive Community-dwelling People Aged ≥65 Years
Brief Title: A RCT Evaluating a Chatbot in Increasing Physical Activity Among Older Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Zixin Wang, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 20210531
Record Dates: First submitted 2024-10-12; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Physical Inactivity
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The Chatbot will assess participants' physical activity level and stage of changes regarding physical activity and automatically deliver interventions tailor to their stage of changes every week for 12 weeks. The Chatbot will address questions related to physical activity raised by the participants.
  Interventions: Behavioral: Chatbot-delivered interventions tailored to one's stage of changes
- Control (Active Comparator): The Chatbot will not assess participants' stage of changes. It will assess participants' physical activity level and provides a standard intervention covering general information about physical activity for older adults, which is not tailoring to participants' stage of changes every week for 12 weeks. The Chatbot will address questions related to physical activity raised by the participants.
  Interventions: Behavioral: Chatbot-delivered standard interventions

INTERVENTIONS:
Behavioral: Chatbot-delivered interventions tailored to one's stage of changes — The Chatbot will assess participants' physical activity level and stage of changes regarding physical activity and automatically deliver interventions tailor to their stage of changes every week for 12 weeks. The Chatbot will address questions related to physical activity raised by the participants.
  Arms: Intervention
Behavioral: Chatbot-delivered standard interventions — The Chatbot will not assess participants' stage of changes. It will assess participants' physical activity level and provides a standard intervention covering general information about physical activity for older adults, which is not tailoring to participants' stage of changes every week for 12 weeks. The Chatbot will address questions related to physical activity raised by the participants.
  Arms: Control

SUMMARY:
This study will compare the efficacy of a Chatbot-delivered stage of changes (SOC)-tailored online intervention (intervention group) versus a Chatbot-delivered non-SOC-tailored online intervention in increasing the prevalence of meeting WHO recommended physical activity level six months after completion of the intervention among inactive community-dwelling individuals aged ≥65 yeas. In the intervention group, the Chatbot will assess participants' physical activity level and SOC regarding PA and automatically deliver interventions tailor to their SOC every week for 12 weeks. In the control group, the Chatbot will not assess participants' SOC. It will assess participants' physical activity level and provides a standard intervention covering general information about physical activity for older adults, which is not tailoring to participants'SOC every week for 12 weeks. All participants will be followed up after completion of the interventions (T1) and six months after T1 (T2).

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥65 years,
* Having a Hong Kong ID,
* Chinese speaking,
* Not meet the WHO recommended level of MVPA
* Willing to be followed by telephone at 3 and 9 months,
* Having a smartphone
* Able to send and read text/voice message via smartphone.
* Willing to wear an accelerometer for a week at T0, T1 and T2.

Exclusion Criteria:

* Blindness or deafness,
* Having been diagnosed with major psychiatric illness (schizophrenia or bipolar disorder) or dementia,
* Score ≥1 in the Chinese version of the Physical Activity Readiness Questionnaire (PAR-Q)
* Score ≤16 in the validated telephone version of the Cantonese Mini-mental State Examination (T-CMMSE)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 278 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Meeting WHO recommended level of physical activity | 9 months
  Prevalence of meeting WHO recommended level of physical activity (at least 150 minutes moderate-intensity aerobic physical activity every week) at T1 (after completion of intervention) and T2 (6 months after T1). Physical activity will be measured by self-reported data and using an accelerometer.

CONTACTS AND LOCATIONS:
Overall Officials: Zixin Wang, Dr., Principal Investigator — Centre for Health Behaviours Research, the Chinese University of Hong Kong
Locations (1):
- Centre for Health Behaviours Research, the Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liang X, Sun F, Zhang Q, Fang Y, Yu FY, Ye D, Zhang B, Liao Q, Mo PK, Wang Z. Chatbot-Delivered Stage of Change-Tailored Web-Based Intervention to Promote Physical Activity Among Inactive Community-Dwelling People Aged 65 years or More: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Jun 20;14:e68796. doi: 10.2196/68796. PMID 40540737